CLINICAL TRIAL: NCT02280291
Title: Comparison Between Single Shot Peripheral Nerve Block and Continuous Infusion Via a On-Q Pump in Extremity Fracture Operations: a Randomized Prospective Control Trial
Brief Title: Single Shot Versus OnQ Pump in Extremity Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-03598
Record Dates: First submitted 2014-10-15; First posted 2014-10-31 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Pain; Fracture
MeSH Terms: conditions — Pain; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ankle Single Shot Block (SSB) (Active Comparator)
  Interventions: Drug: Ankle SSB
- Ankle OnQ (Continuos Sedation OnQ Pump) (Experimental)
  Interventions: Drug: Ankle OnQ
- DR SSB (Experimental)
  Interventions: Drug: DR SSB
- DR OnQ (Experimental)
  Interventions: Drug: DR OnQ

INTERVENTIONS:
Drug: Ankle SSB — general anesthesia/sedation with a single shot; Primary predictor variable: single shot block, a 22 gauge, 3.5 inch needle will be used and 20cc of 2% lidocaine with 1:200,000 epinephrine + 20cc of 0.5% bupivacaine with 1:300,000 epinephrine will be injected around the nerve after confirming negative aspiration every 5 cc.
  Arms: Ankle Single Shot Block (SSB)
Drug: Ankle OnQ — versus regional block with continuous infusion using an OnQ pump. 17 gauge Tuohy needle will be used and 20cc of 2% lidocaine with epinephrine +20cc of 0.5% bupivacaine with1:300,000epinephrine will be injected around the nerve after confirming negative aspiration every 5cc.
  Arms: Ankle OnQ (Continuos Sedation OnQ Pump)
Drug: DR SSB — general anesthesia/sedationwith a single shot; general anesthesia/sedation with a single shot; Primary predictor variable: single shot block, a 22 gauge, 3.5 inch needle will be used and 20cc of 2% lidocaine with 1:200,000 epinephrine + 20cc of 0.5% bupivacaine with 1:300,000 epinephrine will be injected around the nerve after confirming negative aspiration every 5 cc.
  Arms: DR SSB
Drug: DR OnQ — versus regional block with continuous infusion using an OnQ pump. 17 gauge Tuohy needle will be used and 20cc of 2% lidocaine with epinephrine +20cc of 0.5% bupivacaine with1:300,000epinephrine will be injected around the nerve after confirming negative aspiration every 5cc.
  Arms: DR OnQ

SUMMARY:
Peripheral nerve blocks have been well studied in the literature with generally good results for controlling post operative pain following orthopaedic surgery. Regional anesthesia has many benefits. It provides excellent intraoperative anesthesia and muscle relaxation as well as analgesia that continues into the post-operative period. These regional blocks are also effective in controlling pain in the immediate post-operative period. However, as the block wears off, patients begin experiencing increased pain. Compared to patients treated without regional blocks, these patients will often experience a "rebound pain"--pain occurring 12-24 hours after surgery that is subjectively worse than that in patients treated without regional blocks. Therefore, the investigators propose to use a continuous infusion of anesthetic in order to provide sustained pain control post-operatively. Preoperatively, patients will be randomized into a single shot peripheral nerve block versus a continuous infusion of peripheral nerve block. Post-operatively, pain will be assessed using the Visual Analogue Scale (1-100) prior to being discharged from PACU. Time to discharge and amount of pain medication taken will be recorded. Patients will be contacted at certain time intervals postoperatively to assess their pain scale and pain medication intake. Patients will be seen for routine post-operative follow-up visits where they will be assessed for satisfaction, pain, residual neurological symptoms, and signs of infection.

DETAILED DESCRIPTION:
Purpose The purpose of this randomized prospective study will be to compare post-operative pain control after extremity fracture fixation surgery between patients who receive single shot versus continuous peripheral nerve blocks.

Scientific or Scholarly Rationale Peripheral nerve blocks have been well studied in the literature with generally good results for controlling post operative pain following orthopaedic surgery 1-4. Regional anesthesia has many benefits. It provides excellent intraoperative anesthesia and muscle relaxation as well as analgesia that continues into the post-operative period. Airway manipulations are avoided, post-operative nausea and vomiting are diminished, post-anesthesia care unit stay are shortened, and fewer nursing interventions in the post-anesthesia care unit are required5-6.

Patients who have operative fixation of extremity fractures (ankle, wrist, forearm) are typically ambulatory patients. However, many become hospitalized overnight secondary to inadequate pain control, increasing hospital costs. Goldstein et al. showed that patients who underwent popliteal blocks after ankle fracture fixation demonstrated significantly better pain control immediately postoperatively7. The need for overnight hospitalization secondary to pain is decreased, as are nonsurgical operating room times.

Despite the success of regional anesthesia, a phenomenon known as "rebound pain" has been shown to occur as the original block wears off7-9. Patients with blocks will experience significantly increased pain compared to those without blocks approximately 12-24 hours after surgery. This can be controlled with early narcotic administration but can be a source of significant discomfort to a patient if not recognized and treated in time. A few studies have shown that continuous infusions of various numbing agents are efficacious in prolonged pain control, even in the ambulatory setting10-12. Nevertheless, no studies have thus performed a randomized prospective control trial studying the efficacy of continuous infusion therapy on pain control following extremity fracture surgery.

Aims

1. To determine the effectiveness of continuously infused regional anesthetic for pain control in extremity fracture surgery
2. To determine the effect of rebound pain on patient satisfaction of surgery Description of study and study procedure Consent All patients being treated with open reduction internal fixation for foot, ankle, tibia, elbow, forearm and wrist fractures at New York University Medical Center, NYU-Hospital for Joint Diseases will be asked to participate in this study. At the patients preoperative office visit, they will be asked to participate in the study and provided a copy of the consent form at that time which they can take home with them. All questions will be answered and they will be asked verbally if they will consent to being a part of the study. Patients will then have the opportunity to either sign the written consent forms or wait till the surgical date to think about the study and any additional questions they may have. At the time of surgery, patients will be consented for surgery. If the patient did not give written consent at the preoperative visit, they will be asked if they have any questions about the study. All questions will again be answered. They will then be asked verbally if they are willing to participate in the study, if they respond yes, then written consent will be obtained at that time.

Randomization Patients will then be randomized (using an online randomizer, similar to a flip of a coin) to one of two anesthetic protocols: regional block with single dose of anesthetic versus regional block with continuous infusion using an OnQ pump. If for some reason, the anesthesiologist feels that a patient would benefit from one type of anesthesia over another, the patient will be removed from the study and given that type of anesthesia.

Intervention Patients will be randomized to one of two anesthetic protocols: general anesthesia/sedation with a single shot, peripheral nerve block versus general anesthesia/sedation with a continuous, peripheral nerve block.

All anesthesia will be provided by an attending anesthesiologist with or without an anesthesiology resident/CRNA. Patients will have standard ASA monitors placed (pulse oximeter, blood pressure, EKG) and an intravenous line started. Sedation will be given using a combination of midazolam (1-4 mg) and fentanyl (25-100 mcg). Patients in both groups will receive an ultrasound-guided peripheral nerve block. The block will be either an infraclavicular brachial plexus block or a popliteal nerve block, depending on the location of the fracture. The appropriate region will be prepped with a chlorohexidine solution on the appropriate surgical side and the appropriate site will be visualized under ultrasound. For the group receiving a single shot block, a 22 gauge, 3.5 inch needle will be used and 20cc of 2% lidocaine with 1:200,000 epinephrine + 20 cc of 0.5% bupivacaine with 1:300,000 epinephrine will be injected around the nerve after confirming negative aspiration every 5 cc. For those receiving a continuous infusion, a 17 gauge Tuohy needle will be used and 20cc of 2% lidocaine with epinephrine + 20 cc of 0.5% bupivacaine with 1:300,000 epinephrine will be injected around the nerve after confirming negative aspiration every 5cc. Once the injection is complete, an indwelling catheter will be placed with its tip location confirmed and then secured at the skin.

After placement of the regional block, general anesthesia/sedation will be administered and maintained at the discretion of the anesthesiologist. Induction of anesthesia will involve IV propofol (2mg/kg) and fentanyl (1-2mcg/kg). Neuromuscular blockade will be used at the discretion of the anesthesiologist and will be reversed appropriately. Anesthetic maintenance will involve inhalational agents, IV agents, air, and oxygen. Fentanyl will be the only intraoperative analgesic used and will be dosed as determined by the anesthesiologist.

After completion of the surgery, patients will be taken to the PACU where those with continuous catheters will have an OnQ pump attached to it. The patient will begin receiving a continuous infusion of 0.2% ropivacaine through the catheter at a rate of 8 cc/hr. The patient will be discharged home with the catheter for 48 hours. The study participant will self-discontinue the catheter in 2 days. This involves removing the tegaderm dressing and gently pulling the catheter out from under the skin. A bandage may then be applied. Germaine Cuff, the investigators anesthesiology RN, will be available via phone to answer any questions study participants may have regarding discontinuation of the catheter. Breakthrough pain while in the PACU will be treated with IV fentanyl and PO Percocet as needed.

Postoperatively, all patients will be discharged home with a prescription for Percocet 5/325 with instructions to take 1-2 tabs every 4-6hrs as needed for pain.

Data collection Location and type of surgical procedure, duration of procedure, and duration of intravenous sedation will also be recorded. Total time in the operating room will also be noted. Time admitted to PACU, time clinically ready for discharge, time actually discharge, PACU medications for nausea/vomiting and PACU meds for pain will all be recorded prior to discharge.

Post-operative pain will be assessed using the Visual Analogue Scale (0-100) prior to being discharged from PACU. Time to discharge and amount of pain medication taken in the PACU will be recorded.

Patients will be contacted 8 hours, 12 hours, 24 hours, 48 hours and 72hrs after surgery by the operative surgeon or research coordinator to assess their pain scale and pain medication intake. Patients will be seen for routine post-operative follow-up visits at two, six, twelve, twenty-four, and fifty-two weeks. At these times, patients will be assessed for pain, residual neurological symptoms, and signs of infection. Patients will also be asked if they were satisfied with their postoperative pain control. Total duration of study will be fifty-two weeks. Data collection documents will be distributed to the patients at time of surgery to assist in patient understanding.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at least 18 years old.
2. Male or Female
3. All racial and ethnic groups
4. Fractures and fracture/dislocations of the foot, ankle, tibia, fibula, elbow, forearm, wrist and hand
5. Patients who opt for surgical treatment of their fractures.
6. Patients who consent to be randomized.
7. Patients who are willing to follow-up for a minimum of 52 weeks.

Exclusion Criteria:

1. Patients younger than 18 years old.
2. Patients who are on chronic opioids
3. Patients who abuse opioids
4. Patients who are unwilling to follow-up for a minimum of 52 weeks.
5. Neurologic condition that could interfere with pain sensation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirmal Tejwani, MD, Principal Investigator — NYU Hospital for Joint Diseases
Locations (1):
- Hospital for Joint Diseases, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ankle Single Shot Block (SSB) | Ankle OnQ (Continuos Sedation OnQ Pump) | DR SSB | DR OnQ
Started | 25 | 25 | 24 | 26
Completed | 21 | 23 | 21 | 18
Not Completed | 4 | 2 | 3 | 8
Not completed — Lost to Follow-up | 2 | 1 | 3 | 8
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ankle Single Shot Block (SSB) | Ankle OnQ (Continuos Sedation OnQ Pump) | DR SSB | DR OnQ | Total
Number analyzed (Participants) | 25 | 25 | 24 | 26 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 21 | 20 | 20 | 83
  >=65 years | 3 | 4 | 4 | 6 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 17 | 16 | 59
  Male | 10 | 14 | 7 | 10 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 17 | 16 | 59
  Male | 10 | 14 | 7 | 10 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 24 | 26 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on Visual Analog Scale (VAS)
Description: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 ("no pain") and 10 ("worst pain").
Time Frame: 2 weeks, 6 weeks
Population: Some of the number of participants analyzed differs from the overall number analyzed because some participants were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ankle Single Shot Block (SSB) | Ankle OnQ (Continuos Sedation OnQ Pump) | DR SSB | DR OnQ
Number analyzed (Participants) | 20 | 23 | 13 | 12
score on a scale
  2 weeks post-op: number analyzed (Participants) | 17 | 23 | 13 | 12
  2 weeks post-op | 3.28 (2.26) | 1.47 (1.42) | 3.62 (1.71) | 3.91 (3.12)
  6 weeks post-op: number analyzed (Participants) | 20 | 21 | 13 | 11
  6 weeks post-op | 1.8 (2.53) | 0.62 (0.98) | 3.46 (2.96) | 2.58 (2.91)

2. Secondary Outcome: Disability of the Arm, Shoulder and Hand (DASH) Score
Description: The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Time Frame: 2 Weeks, 6 Weeks
Population: Data was not collected for the Ankle SSB and Ankle OnQ arms, as the DASH scale is upper extremity-specific (including only arm, shoulder, and hand disabilities).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DR SSB | DR OnQ
Number analyzed (Participants) | 13 | 12
score on a scale
  2 weeks | 53.97 (18.56) | 62.17 (19.94)
  6 weeks | 36.78 (25.77) | 45.69 (32.36)

ADVERSE EVENTS:
Time Frame: 6 Weeks Post Op
Arm/Group | Ankle Single Shot Block (SSB) | Ankle OnQ (Continuos Sedation OnQ Pump) | DR SSB | DR OnQ
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/24 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT02280291/Prot_SAP_000.pdf